CLINICAL TRIAL: NCT03190863
Title: Investigating the Effect of Motor Imagery With or With no Visual Neurofeedback on Grasping Capabilities After C6-C7 Tetraplegia: a Multicentric Randomized Controlled Trial.
Brief Title: Grasping Rehabilitation Using Motor Imagery With or With no Neurofeedback After Tetraplegia
Acronym: TETRAMINF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 69HCL17_0016
Record Dates: First submitted 2017-04-25; First posted 2017-06-19 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Individuals With C6-C7 Tetraplegia (AIS A or B)
Keywords: Tenodesis grasp; Neurofeedback; Motor imagery; Reach-to-grasp; Rehabilitation; Physical therapy; Cervical spinal cord injury; Tetraplegia; AIS A; AIS B
MeSH Terms: conditions — Quadriplegia | interventions — Neurofeedback

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motor imagery combined with neurofeedback (MINF) (Experimental)
  Interventions: Behavioral: Motor imagery combined with neurofeedback (MINF)
- Motor imagery (MI) (Active Comparator)
  Interventions: Behavioral: Motor imagery (MI)
- Control (C) (Sham Comparator)
  Interventions: Behavioral: Control (C)

INTERVENTIONS:
Behavioral: Motor imagery combined with neurofeedback (MINF) — 7 individuals with C6-C7 tetraplegia randomize in the experimental group consisting in motor imagery practice combined with visual neurofeedback (NF - i.e. performance of the imagined movement).
  Intervention consists in a total of 15 sessions repeated 3 times a week and lasting 5 weeks. Each session will last 45 minutes. An experienced physical therapist supervised all sessions. After each imagined movement, the NF based on brain activity measured by electroencephalography is display on a screen.
  Arms: Motor imagery combined with neurofeedback (MINF)
Behavioral: Motor imagery (MI) — 7 individuals with C6-C7 tetraplegia randomized in the active comparator group consisting in motor imagery practice alone without visual NF. This means that the performance of the imagined movement is not displayed to the participants.
  Intervention consists in a total of 15 sessions repeated 3 times a week and lasting 5 weeks. Each session will last 45 minutes. An experienced physical therapist supervised all sessions.
  Arms: Motor imagery (MI)
Behavioral: Control (C) — 7 individuals with C6-C7 tetraplegia randomized in the sham comparator group consisting in imagining geometric shapes by visualization. Shapes are successively displayed on a screen.
  Intervention consists in a total of 15 sessions repeated 3 times a week and lasting 5 weeks. Each session will last 45 minutes. An experienced physical therapist supervised all sessions.
  Arms: Control (C)

SUMMARY:
Motor imagery has shown promising results to optimize tenodesis grasp in individuals with C6-C7 tetraplegia. However, efficacy of using motor imagery to improve grasping after tetraplegia requires further study with higher level of evidence. In addition, controlling covert practice remains difficult due to the absence of overt movements. However, similar brain activity measured during both over and cover movements makes possible to provide visual information about the covert practice performance using neurofeedback.

The Investigators thus designed this multicentric randomized controlled trial to investigate the effect of motor imagery with or with no visual neurofeedback on grasping capabilities after C6-C7 tetraplegia. They hypothesized that providing neurofeedback based on brain activity measured by electroencephalography namely knowing the covert practice performance would results in greater grasping improvement in response to practice as compared to motor imagery practice alone.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer individuals with C6-C7 tetraplegia with complete finger flexor paralysis restricting grasping capabilities to the tenodesis.
* Consent to participate to the study after receiving clear, loyal and appropriate information.
* Aged between 18 and 55 years.
* Time since spinal cord injury above 6 months
* Stabilized condition in particular sensori-motor deficit.
* Sitting position for more than 1 hour
* Able to imagine movement
* Health care beneficiary

Exclusion Criteria:

* Long-lasting autonomic disorders while sitting (orthostatic hypotension and/or blood pressure instability) limiting sitting position to less than 1 hour.
* Upper limb pain for either mechanic or neuropathic reasons preventing all grasping movement and/or the ability to imagine those movements.
* Restricted wrist and finger range of motion preventing the tenodesis grasp.
* Patient after surgical tendon transfer that improved grasping capabilities (e.g. active finger flexion).
* Ongoing participation in another research that aim to evaluate an intervention likely to improve the neurological or functional recovery introducing an experimental bias.
* Specific contraindication to Magnetoencephalography with the presence of metallic fragments inside the body such as pace-maker, neurostimulator, cochlear implants, steel dental implant and osteosynthesis material only applicable to the participants included in Lyon hospital center (n=15).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2018-03-29 (Actual); Primary Completion 2025-05-29 (Estimated); Study Completion 2025-05-29 (Estimated)

PRIMARY OUTCOMES:
Wrist extension angle in degree during grasping with 3D motion analysis system | Up to 19 weeks
  Individuals with C6-C7 tetraplegia extend their wrist to grasp using tenodesis. Specifically, the wrist extension shortens the tendons of fingers and thumbs flexors that elicit either a palmar or a lateral grip. A complete reach-to-grasp movement will be recorded using a 3D motion analysis system (Vicon Motion Systems Ltd. UK). Wrist extension angle in degree will be measure during grasping when the object is grasped.

SECONDARY OUTCOMES:
Temporal kinematic parameters of reach-to-grasp movements with 3D motion analysis system (Vicon Motion Systems Ltd. UK). | Up to 19 weeks
  Computation of temporal kinematic parameters (e.g. movement duration) measured during a complete reach-to-grasp movement using a 3D motion analysis system (Vicon Motion Systems Ltd. UK). Temporal parameters are also aggregated with spatial parameters.
Spatial kinematic parameters of reach-to-grasp movements with 3D motion analysis system (Vicon Motion Systems Ltd. UK). | Up to 19 weeks
  Computation of spatial kinematic parameters (e.g. movement trajectory) measured during a complete reach-to-grasp movement using a 3D motion analysis system (Vicon Motion Systems Ltd. UK).Spatial parameters are also aggregated with temporal parameters.
Brain activity change in response to intervention using magnetoencephalography | Up to 19 weeks
  Brain activity will be measured during upper limb movement (e.g. a complete reach-to-grasp movement) using magnetoencephalography. The device is only available in Lyon Hospital. Correspondingly, fifteen participants included in Lyon Hospital will achieve this measure.
passive upper limb range of motion (ROM) measured using goniometer and/or inclinometer | Up to 19 weeks
  This outcome will be measured using goniometer and/or inclinometer by the same blind and experienced physical therapist
Upper limb strength measured using the hand held dynamometer | Up to 19 weeks
  This outcome will be measured using the manual muscle test and the hand held dynamometer by the same blind and experienced physical therapist.
Upper limb strength measured using the manual muscle test | Up to 19 weeks
  This outcome will be measured using the manual muscle test and the hand held dynamometer by the same blind and experienced physical therapist.
Hand dexterity measured using the Box and Block test | Up to 19 weeks
  This outcome will be measured using i) the Box and Block Test, ii) the Nine Hole Peg Test, iii) the Jebsen Test and iv) the Capability of Upper Limb Test supervised by the same blind and experienced occupational therapist
Hand dexterity measured using the Nine Hole Peg test | Up to 19 weeks
  This outcome will be measured using i) the Box and Block Test, ii) the Nine Hole Peg Test, iii) the Jebsen Test and iv) the Capability of Upper Limb Test supervised by the same blind and experienced occupational therapist
Hand dexterity measured using the Jebsen test | Up to 19 weeks
  This outcome will be measured using i) the Box and Block Test, ii) the Nine Hole Peg Test, iii) the Jebsen Test and iv) the Capability of Upper Limb Test supervised by the same blind and experienced occupational therapist
Hand dexterity measured using the Capability of Upper Limb test | Up to 19 weeks
  This outcome will be measured using i) the Box and Block Test, ii) the Nine Hole Peg Test, iii) the Jebsen Test and iv) the Capability of Upper Limb Test supervised by the same blind and experienced occupational therapist
Quality of Life measured using the WHOQOL-Bref | Up to 19 weeks
  This outcome will be measured using the WHOQOL-Bref by the same blind and experienced physical therapist.
Daily life autonomy measured using the Quadriplegic Index of Function | Up to 19 weeks
  This outcome will be measured using the Quadriplegic Index of Function by the same blind and experienced physical therapist.
Motor imagery capability measured by the Kinesthetic Visual Imagery Questionnaire | Up to 19 weeks
  Motor imagery capability will be measured by the Kinesthetic Visual Imagery Questionnaire by the same blind and experienced physical therapist along with comparing overt and covert movement duration, galvanic skin response, electroencephalography activity.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien MATEO, PhD, Principal Investigator — Hospices Civils de Lyon, Hôpital Henry Gabrielle, Plate-forme Mouvement et Handicap, F-69000 Lyon, France.
Locations (2):
- France (2):
  - Le Centre Mutualiste Neurologique PROPARA, Parc Euromédecine, Montpellier
  - Service de médecine physique et de réadaptation, Hôpital Henry Gabrielle, Saint-Genis-Laval

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared after deidentification (but only the data required for the new analysis will be transmitted). This includes for each visit and each participant averaged data of wrist extension angle during grasping of a single upper limb measured in degree with 3D motion analysis system.
  This includes for each visit, each participant and each upper limb:
  * Box and Block test
  * Nine Hole Peg test
  * hand held dynamometer for each of 4 muscles
  This includes for each visit and each participant the total score of:
  * manual muscle testing of the upper limb key muscles as defined by the ASIA score for each arm
  * Capability of Upper Limb
  * WHOQOL-Bref
  * Quadriplegic Index of Function
  * Kinesthetic Visual Imagery Questionnaire This also includes for each visit and each participant the passive range of motion expressed in degree and measured using goniometer for shoulder, elbow and wrist.
  This do not include electrophysiological measurements.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Immediately following publication and ending 5 years following article publication.
Access Criteria: Proposals should be directed to sebastien.mateo@chu-lyon.fr. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Mateo S, Di Rienzo F, Reilly KT, Revol P, Delpuech C, Daligault S, Guillot A, Jacquin-Courtois S, Luaute J, Rossetti Y, Collet C, Rode G. Improvement of grasping after motor imagery in C6-C7 tetraplegia: A kinematic and MEG pilot study. Restor Neurol Neurosci. 2015;33(4):543-55. doi: 10.3233/RNN-140466. PMID 26409412
- [Derived] Charbonnier G, Reilly KT, Schwartz D, Daligault S, Luaute J, Rossetti Y, Collet C, Gelis A, Rode G, Mateo S. Grasping rehabilitation using motor imagery with or without neurofeedback after tetraplegia: a study protocol for a bicentric randomised controlled trial. BMJ Open. 2024 Oct 21;14(10):e074652. doi: 10.1136/bmjopen-2023-074652. PMID 39433413